CLINICAL TRIAL: NCT04611568
Title: Educational Program for the Early Detection of Melanoma in Oregon
Brief Title: War on Melanoma™ Public Health & Education Campaign
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Melanoma Research Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Sancy A Leachman, MD, PhD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00019372; NCI-2020-01301 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019372 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (health educational campaign) (Experimental): MEDIA CAMPAIGN: Participants view digital media strategies.
  PRIMARY CARE PROVIDERS AND PROFESSIONALS: Primary care providers and professionals who see skin and potential melanomas receive online based curriculum on melanoma. Participants also complete a survey to assess knowledge and confidence before and after receiving the curriculum.
  MELANOMA COMMUNITY REGISTRY VOLUNTEERS: Melanoma Community Registry volunteers in Oregon receive educational and training materials on melanoma. Participants also complete a survey before and after receiving educational material.
  HIGH SCHOOL STUDENTS: High school students receive an educational lecture over 1 hour on sun-safety and early detection of melanoma practices. Participants also complete a survey before and after the educational lecture.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Behavioral: Media Campaign; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational and training material
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Educational Intervention — Receive educational lecture
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Health Education — Receive melanoma curriculum
Behavioral: Media Campaign — View digital media strategies
Other: Survey Administration — Complete survey

SUMMARY:
This trial studies how well a health educational campaign works in increasing early detection of melanoma in Oregon. The health educational campaign may provide information to help people learn about the early signs of melanoma. Increased education in Oregon may decrease the number of people who die from melanoma and increase the number of melanomas that are identified at an earlier stage.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the change in melanoma literacy in Oregon, Washington, and Utah over five years (relative to baseline) and determine if there is a statistically significant difference in literacy in Oregon (where the educational campaign occurred) as compared to the non-participating states (Washington and Utah).

II. To determine if there is an association between melanoma literacy and 1) stage at diagnosis, 2) tumor depth, 3) incidence, and 4) mortality rates in Oregon, Washington, and Utah.

III. To determine if the cost of care for melanoma in Oregon is impacted by melanoma literacy and/or tumor stage.

OUTLINE:

MEDIA CAMPAIGN: Participants view digital media strategies.

PRIMARY CARE PROVIDERS AND PROFESSIONALS: Primary care providers and professionals who see skin and potential melanomas receive online based curriculum on melanoma. Participants also complete a survey to assess knowledge and confidence before and after receiving the curriculum.

MELANOMA COMMUNITY REGISTRY VOLUNTEERS: Melanoma Community Registry volunteers in Oregon receive educational and training materials on melanoma. Participants also complete a survey before and after receiving educational material.

HIGH SCHOOL STUDENTS: High school students receive an educational lecture over 1 hour on sun-safety and early detection of melanoma practices. Participants also complete a survey before and after the educational lecture.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, melanoma patients, skin service providers and health care providers interested in awareness and educational campaign

Exclusion Criteria:

* No one will be intentionally excluded

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75000 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Statewide awareness (level of knowledge and detection) | Up to completion of surveys, assessed up to 5 years
  Will compare the level of knowledge and early detection of melanoma between participants in Oregon who received the educational campaign and those who did not in Washington and Utah.
Cancer data collection (correlation with demographic and geographic factors) | Up to 5 years
  Will collect baseline and post-intervention data from Oregon State Cancer Registry (OSCaR) on melanoma diagnoses to correlate the incidence and pathologic factors with demographic and geographic factors.
Cost data | Up to 5 years
  Will compare reports of cost data between those who received the health education campaign and those who did not.
Reach of educational campaign | Up to completion of surveys, assessed up to 5 years
  Will determine the reach of the educational campaign across Oregon using volunteer activity logs, volunteer training logs, and website usage analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sancy A Leachman, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- See also: Web site describing the project. — http://www.WarOnMelanoma.org
- See also: Unbranded Early Detection Campaign — http://www.StartSeeingMelanoma.com